CLINICAL TRIAL: NCT01140243
Title: Efficacy and Suitability of Infant Formula With a Special Fat Formulation for Premature Infants Following Discharge From Hospital Following Discharge From Hospital
Brief Title: Infant Formula Supplemented With a Special Fat Formulation for Premature Infants Following Discharge From Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Materna Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 030
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2012-04

CONDITIONS: Premature Infants
Keywords: fat formulation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test product (Experimental): Dietary supplement
  Interventions: Dietary Supplement: LCPUFA
- standart (Active Comparator): Dietary supplement
  Interventions: Dietary Supplement: LCPUFA

INTERVENTIONS:
Dietary Supplement: LCPUFA — premature infant formula supplemented with LCPUFA

SUMMARY:
The purpose of this study is to compare the efficacy and nutritional suitability of 2 infant formulas supplemented with different levels of LCPUFA, for premature infants following discharge from Hospital.

ELIGIBILITY:
Inclusion Criteria:

* premature infants of gestational age 32-34 weeks and AGA birth weight who are healthy at time of discharge.
* whose mothers are unable to breast feed or have chosen not to breast feed,
* Whose parents have signed the informed consent form.
* Only the first among twins will be recorded for the study.

Exclusion Criteria:

* Chromosomal abnormalities or congenital malformation.
* Metabolic abnormalities.
* Central nervous system abnormalities.
* Severe developmental disorders.
* GI problems, GI surgery, necrotizing enterocolitis (NEC), gastro-esophageal reflux disease (GERD) requiring nutritional intervention.
* Milk allergy or intolerance.
* Growth failure.
* Chronic disease

Ages: 2 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
anthropometric | 12 weeks
  anthropometric measure will be taken at the time of recruitment and on the following 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Neonatal Intensive Care Unit, Barzilai Medical Center, Ashkelon
  - Sharei Zedek MC, Jerusalem